CLINICAL TRIAL: NCT06177418
Title: Glove Finger Method to Prevent Wound Infection in Children Undergoing Transumbilical Laparoscopic Appendectomy
Brief Title: Transumbilical Laparoscopic Appendectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmi Kadıoğlu Hospital (Other)
Responsible Party: Principal Investigator, Mustafa Azizoğlu, Medical Doctor, Necmi Kadıoğlu Hospital, Necmi Kadıoğlu Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2023-12-10; First posted 2023-12-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Appendicitis; Surgical Site Infection
Keywords: laparoscopic appendectomy; transumbilical laparoscopic appendectomy; appendicitis; children; surgical site infection
MeSH Terms: conditions — Appendicitis; Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard transumbilical laparoscopic appendectomy (Active Comparator): In this group, patients will undergo the standard transumbilical laparoscopic appendectomy procedure through a 15 mm trocar port in the umbilical region. The procedure will involve locating the appendix and removing it via an extracorporeal approach.
  Interventions: Procedure: Standard transumbilical laparoscopic appendectomy
- Transumbilical laparoscopic appendectomy + glove finger technique (Experimental): In addition to the standard transumbilical laparoscopic appendectomy procedure, patients in this group will receive the glove finger technique, aimed at preventing contamination of surrounding tissues by infected tissue.
  Interventions: Procedure: Transumbilical laparoscopic appendectomy + Glove finger technique

INTERVENTIONS:
Procedure: Transumbilical laparoscopic appendectomy + Glove finger technique — Ssince the appendix becomes infected when it is removed from the umbilicus, the infected appendix contacts the edge of the incision during release, thus contaminating the incision and causing postoperative wound infection. Additionally, in the experimental, to prevent this wound infection, after the appendix is taken out through the umbilical incision, the appendix is placed inside the glove finger, thus preventing the appendix from touching the wound during its release. This reduces wound infection in the postoperative period.
  Arms: Transumbilical laparoscopic appendectomy + glove finger technique
Procedure: Standard transumbilical laparoscopic appendectomy — Standart transumbilical laparoscopic appendectomy
  Arms: Standard transumbilical laparoscopic appendectomy

SUMMARY:
Transumbilical laparoscopic appendectomy (TULA) is increasingly favored in the treatment of appendicitis within the realm of minimally invasive surgical approaches. This procedure offers advantages such as superior cosmetic outcomes and reduced postoperative pain. However, like all surgical interventions, it carries the inherent risk of surgical site infections (SSI), which pose significant challenges to patient health and healthcare systems by escalating treatment costs, prolonging recovery, and increasing morbidity rates. This study aims to evaluate the efficacy of the "glove finger method" in mitigating SSI risk in TULA.

The rationale for this study is predicated on the hypothesis that the glove finger method could serve as a simple and cost-effective measure offering potential protection against SSIs. When compared to traditional methods, this technique may not only reduce surgical duration but also diminish the risk of SSIs, thereby potentially decreasing hospital stay durations. Furthermore, enhancing the understanding of factors contributing to the development of SSIs and developing effective strategies for their prevention can elevate patient care quality and alleviate the burden on healthcare systems.

DETAILED DESCRIPTION:
Transumbilical laparoscopic appendectomy (TULA) is increasingly favored in the treatment of appendicitis within the realm of minimally invasive surgical approaches. This procedure offers advantages such as superior cosmetic outcomes and reduced postoperative pain. However, like all surgical interventions, it carries the inherent risk of surgical site infections (SSI), which pose significant challenges to patient health and healthcare systems by escalating treatment costs, prolonging recovery, and increasing morbidity rates. This study aims to evaluate the efficacy of the "glove finger method" in mitigating SSI risk in TULA.

The rationale for this study is predicated on the hypothesis that the glove finger method could serve as a simple and cost-effective measure offering potential protection against SSIs. When compared to traditional methods, this technique may not only reduce surgical duration but also diminish the risk of SSIs, thereby potentially decreasing hospital stay durations. Furthermore, enhancing the understanding of factors contributing to the development of SSIs and developing effective strategies for their prevention can elevate patient care quality and alleviate the burden on healthcare systems.

This study will compare transumbilical laparoscopic appendectomy (TULA) methods applied to pediatric patients diagnosed with acute appendicitis at our clinic. Employing a randomized controlled design, the study aims to assess the efficacy and safety differences between two distinct surgical techniques currently in practice.

The study will adopt a randomized, controlled, and prospective design. Patients will be randomly allocated into two groups based on the treatment methods:

Group 1: Standard TULA Group: In this group, patients will undergo the standard TULA procedure through a 15 mm trocar port in the umbilical region. The procedure will involve locating the appendix and removing it via an extracorporeal approach.

Group 2: TULA + Glove Finger Technique Group: In addition to the standard TULA procedure, patients in this group will receive the glove finger technique, aimed at preventing contamination of surrounding tissues by infected tissue.

The research will examine parameters such as age, gender, duration of symptoms, laboratory and radiological findings, applied treatment methods, surgical techniques, complications, operation time, and the frequency of postoperative wound infections in both groups. This study intends to shed light on the clinical outcomes of various TULA methodologies.

ELIGIBILITY:
Inclusion Criteria:

patients undergo appendectomy between 5 and 18 years.

Exclusion Criteria:

Comorbidity previous surgery

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-25 (Actual); Primary Completion 2024-09-29 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Operative time | intraopertaive period
  operative time
Postoperative wound infection | 2 weeks
  Postoperative wound infection

CONTACTS AND LOCATIONS:
Locations (1):
- Mustafa Azizoğlu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No